CLINICAL TRIAL: NCT02666716
Title: Pharmacokinetics of Fluconazole Given Intravenously as Prophylaxis or Therapy to Patients With an Invasive Fungal Infection in the Intensive Care Unit (PACIFIC)
Brief Title: Pharmacokinetics of Fluconazole IV as Prophylaxis or Therapy to ICU Patients
Acronym: PACIFIC
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCN-AKF14.06
Record Dates: First submitted 2015-08-12; First posted 2016-01-28 (Estimated); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Candidiasis
Keywords: pharmacokinetics; fluconazole; invasive fungal infection; candidiasis; intensive care unit
MeSH Terms: conditions — Candidiasis; Invasive Fungal Infections | interventions — Fluconazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples for determination of fluconazole and free fluconazole
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fluconazole — Dose according to summary of product characteristics (SPC) or local protocols
  Other Names: Diflucan

SUMMARY:
The pharmacokinetics of fluconazole are expected to be different in ICU patients compared to non-ICU patients. The investigators will determine fluconazole and free fluconazole concentrations in 20 ICU patients, who will get intravenous fluconazole as standard care. Switching to oral/enteral fluconazol is allowed after day 3.

A full pharmacokinetic curve will be taken on day 3 of iv therapy and limited pharmacokinetic curves on day 7 of iv therapy and/or on day 3 of oral therapy; trough levels will be taken daily after intravenous therapy.

DETAILED DESCRIPTION:
The pharmacokinetics of fluconazole are expected to be different in ICU patients compared to non-ICU patients and healthy volunteers due to underlying disease(s). Therefore, extrapolation of data from healthy volunteers and non-ICU patients is not possible.

To be able to include 20 patients within the study duration, a multi-centre approach is necessary.

Patients will receive standard care, as stated in the product characteristics or according to local protocols. Blood sampling for pharmacokinetic analysis will be retrieved through a central venous catheter. A maximum of 62 milliliter blood in total will be drawn for this study. Patients will be monitored daily during the treatment period for adverse events of the study drug.

Full pharmacokinetic curves will be taken on day 3 of iv therapy. Limited pharmacokinetic curves will be taken on day 7 of iv therapy. These two moments of pharmacokinetic analysis will enable the determination steady state and enable the determination of intra-individual variability.

As probably not all patients included will be treated with iv fluconazole for 7 days, switching to oral/enteral therapy is allowed after day 3. To assess bioavailability limited pharmacokinetic curves will be taken on day 3 of oral/enteral therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is admitted to an ICU
2. Subject is at least 18 years of age on the day of the first dosing
3. Subject is managed with a central venous or arterial catheter

Exclusion Criteria:

1. Is known to be hypersensitive to azole antifungal agents
2. Documented history of sensitivity to medicinal products or excipients similar to those found in the fluconazole preparation
3. Has previously participated in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients receiving fluconazole as prophylaxis or therapy for an (invasive) fungal infection at the ICU will be included.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Area under the curve | Days 3 and 7
  Full pharmacokinetic curves will be taken op Day 3 and Day 7 (fluconazole).

SECONDARY OUTCOMES:
body weight | Days 3 and 7
  Identifying influence of body weight on the pharmacokinetics of fluconazole.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Brüggemann, PharmD, PhD, Principal Investigator — Radboud University Medical Center
Locations (3):
- Netherlands (3):
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Radboud university medical center, Nijmegen
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Result] Muilwijk EW, de Lange DW, Schouten JA, Wasmann RE, Ter Heine R, Burger DM, Colbers A, Haas PJ, Verweij PE, Pickkers P, Bruggemann RJ. Suboptimal Dosing of Fluconazole in Critically Ill Patients: Time To Rethink Dosing. Antimicrob Agents Chemother. 2020 Sep 21;64(10):e00984-20. doi: 10.1128/AAC.00984-20. Print 2020 Sep 21. PMID 32816723